CLINICAL TRIAL: NCT06248645
Title: Oxygen Therapy As an Acute Treatment for Dystonic And/or Plegic Attacks in Alternating Hemiplegia of Childhood
Brief Title: Oxygen As an Acute Treatment in Alternating Hemiplegia of Childhood
Acronym: OXYTAHANE
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: APHP230673
Record Dates: First submitted 2024-01-31; First posted 2024-02-08 (Actual); Last update posted 2024-09-27 (Actual); Status verified 2024-09

CONDITIONS: Alternating Hemiplegia of Childhood
MeSH Terms: conditions — Alternating hemiplegia of childhood | interventions — Oxygen

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Oxygen followed by placebo (Other): Treatment of each motor attacks by oxygen (gaz) during 15 minutes in the first 5 week-period and placebo (medical air) during 15 minutes in the second 5 week-period.
  Interventions: Drug: Oxygen; Drug: Placebo
- Placebo followed by oxygen (Other): Treatment of each motor attacks by placebo (medical air) during 15 minutes, in the first 5 week-period and oxygen (gaz) during 15 minutes in the second 5 week-period.
  Interventions: Drug: Oxygen; Drug: Placebo

INTERVENTIONS:
Drug: Oxygen — High-flow oxygen (12 L/min) administered with a non-rebreathing facial mask, started as soon as possible after the beginning of the attack and for 15 minutes.
Drug: Placebo — High-flow medical air (12 L/min) administered with a non-rebreathing facial mask, started as soon as possible after the beginning of the attack and for 15 minutes.
  Other Names: médical Air

SUMMARY:
Alternating hemiplegia of childhood (AHC) is a rare early-onset neurodevelopmental encephalopathy frequently caused by mutations in the ATP1A3 gene. It is typically characterized by a variable degree of intellectual disability, motor dysfunction and various paroxysmal events (dystonic and plegic attacks). Dystonic and plegic attacks are very disabling and current treatments are disappointing with limited efficacy and poor tolerability. The investigators recently reported the efficacy of high-flow oxygen administration (100% O2 at a flow rate of 12 L/min) as an acute treatment for the dystonic attacks in a 25-year-old patient suffering from AHC. The aim of the study is to assess the effect of high-flow oxygen administration (against placebo) as an acute treatment of dystonic and plegic attacks. The primary outcome will be the proportion of motor attacks stopped 30 minutes after the beginning of motor symptoms over 5 weeks.

DETAILED DESCRIPTION:
This is a multicenter, randomized, placebo-controlled, double-blind crossover study, with two successive periods of 5 weeks.

Participants will be randomized in a 1:1 ratio to receive one of the two treatment sequences: oxygen followed by placebo or placebo followed by oxygen. The two treatment periods will be separated by a wash-out period of 10 days +/- 4 days.

The placebo will consist in the administration of medical air. The same procedure will be used for both treatments (oxygen and medical air): administration with a flow rate of 12 L/min through a non-rebreathing facial mask using indiscernible bottles.

The treatment will be administered as soon as possible after the beginning of the attack and for 15 minutes. If the attack hasn't stopped 30 minutes after the beginning of motor symptoms, the patients will be allowed to receive their usual acute pharmacological treatment if they (or their caregiver) judge it necessary.

The primary outcome will be the proportion of motor attacks stopped 30 minutes after the beginning of motor symptoms over 5 weeks. The secondary outcomes will be:

1. the median duration of dystonic and plegic attacks over 5 weeks
2. the evaluation of the quality of life for patients (PELHS-QOL-2) and caregivers (adapted from the PELHS-QOL-2) at the end of the 5 weeks of treatment
3. the frequency of motor attacks over 5 weeks
4. the consumption of sedative treatments over 5 weeks (number of doses used)
5. treatment tolerance, in particular mouth and nasal dryness, cutaneous irritation, cough, nasal congestion, nausea, other unexpected side effects
6. the proportion of dystonic and plegic attacks respectively stopped 30 minutes after the beginning of motor symptoms over 5 weeks
7. the number and proportion of treated attacks over 5 weeks
8. the number and proportion of attacks starting less than 2 hours after the end of the previous attack
9. the duration of the first attack for each of the two periods of treatment
10. the perception of patients and caregivers at the end of the 5 weeks of treatment, assessed with recorded interviews

ELIGIBILITY:
Inclusion Criteria:

1. Age > 1 year old
2. Patients able to administrate high-flow oxygen through a non rebreathing facial mask, either alone or with assistance
3. Patients with a diagnosis of AHC caused by ATP1A3 mutations presenting at least one dystonic or plegic attack per week lasting more than 30 minutes
4. Absence of long-term treatment or long-term treatment stable over the last month and during the duration of the trial
5. Patients able to give written informed consent
6. Affiliation to social insurance

Exclusion Criteria:

1. Inability for the patients and/or caregivers to follow the protocol (inability to read or understand the instructions, no access to smartphone or computer to fill the informatics patient's form)
2. Patients with severe or uncontrolled obstructive or restrictive chronic respiratory disease (asthma, COPD, obesity, neuromuscular disease), acute systemic aggression (acute coronary syndrome, stroke, sepsis, head trauma) or congenital cardiopathy with a risk of hypercapnia following oxygen administration
3. Women that are pregnant (a negative pregnancy test is required for inclusion) or breath feeding
4. Patients involved in an other clinical trial

Min Age: 1 Year | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2024-09-16 (Actual); Primary Completion 2025-06 (Estimated); Study Completion 2025-06 (Estimated)

PRIMARY OUTCOMES:
Proportion of motor attacks stopped 30 minutes after the beginning of motor symptoms over 5 weeks. | 5 weeks
  The primary outcome will be the proportion of motor attacks stopped 30 minutes after the beginning of motor symptoms over 5 weeks.

SECONDARY OUTCOMES:
the median duration of dystonic and plegic attacks over 5 weeks | 5 weeks
the evaluation of the quality of life for patients (PELHS-QOL-2 Pediatric Epilepsy Learning Healthcare System Quality of Liferated, from 2 to 8) and caregivers (adapted from the PELHS-QOL-2) at the end of the 5 weeks of treatment | 5 weeks
the frequency of motor attacks over 5 weeks | 5 weeks
the consumption of sedative treatments over 5 weeks (number of doses used) | 5 weeks
treatment tolerance, in particular mouth and nasal dryness, cutaneous irritation, cough, nasal congestion, nausea, other unexpected side effects | 5 weeks
the proportion of dystonic and plegic attacks respectively stopped 30 minutes after the beginning of motor symptoms over 5 weeks | 5 weeks
the number and proportion of attacks starting less than 2 hours after the end of the previous attack | 5 weeks
the duration of the first attack for each of the two periods of treatment | 5 weeks
the perception of patients and caregivers at the end of the 5 weeks of treatment, assessed with recorded interviews | 5 weeks

CONTACTS AND LOCATIONS:
Locations (2):
- France (2):
  - HCL LYON, Lyon
  - Hôpital Pitié Salpêtrière, Paris

IPD SHARING:
Plan to Share IPD: No